CLINICAL TRIAL: NCT03444155
Title: Pilot Study for the Evaluation of the Effectiveness of Natural Versus Synthetic Vitamin B Complexes in Humans.
Brief Title: Natural Versus Synthetic Vitamin B Complexes in Human
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Graz (Other)
Responsible Party: Principal Investigator, Priv.-Doz. Mag. Dr. Willibald Wonisch, Principal Investigator, Medical University of Graz
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: Medical University of Graz
Record Dates: First submitted 2018-01-08; First posted 2018-02-23 (Actual); Results first posted 2021-04-26 (Actual); Last update posted 2021-04-26 (Actual); Status verified 2021-04

CONDITIONS: Healthy; Thiamine and Niacin Deficiency States; Pyridoxine Deficiency; Folic Acid Deficiency Anemia, Dietary; Vitamin B 12 Deficiency; Peroxidase; Defect; Polyphenols; Oxidative Stress; Homocystine; Metabolic Disorder
MeSH Terms: conditions — Vitamin B 6 Deficiency; Vitamin B 12 Deficiency; Metabolic Diseases

STUDY DESIGN:
Intervention Model Description: Vitamin B complex (natural vs. synthetic) administered in capsules each day for 6 weeks - 2 weeks wash-out phase I (2 weeks) - cross-over 6 weeks - wash-out phase II (6 weeks)
Who Masked: Participant, Investigator
Masking Description: Masking was organized and supervised by the randomization person in charge. Group assignment was 1:1 (control vs. verum group) with identical packages for both Vitamin supplements with 126 capsules for each subject per phase. Randomization was done with sealed envelopes.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Natural Panmol-B-Complex first, then synthetic Vitamin B-complex (Active Comparator): Participants first received a Natural Vitamin B-complex, i.e., Panmol-B-Complex - B1 (2.93 mg), B2 (3.98 mg), B3 (29.85 mg), B5 (10.95 mg), B6 (3.38 mg), B7 (0.108 mg), B9 (0.69 mg), B12 (8.85 µg) daily each morning for 6 weeks. After a wash-out period of 2 weeks, they then received a synthetic Vitamin B-complex - B1 (2.93 mg), B2 (3.98 mg), B3 (29.85 mg), B5 (10.95 mg), B6 (3.38 mg), B7 (0.108 mg), B9 (0.69 mg), B12 (8.85 µg) daily each morning for 6 weeks.The study finished after the second wash-out period for another 6 weeks.
  Interventions: Dietary Supplement: Natural Panmol-B-Complex
- Synthetic Vitamin B-complex first, then Natural Panmol-B-Complex (Active Comparator): Participants first received a Synthetic Vitamin B-complex - B1 (2.93 mg), B2 (3.98 mg), B3 (29.85 mg), B5 (10.95 mg), B6 (3.38 mg), B7 (0.108 mg), B9 (0.69 mg), B12 (8.85 µg) daily each morning for 6 weeks. After a wash-out period of 2 weeks, they then received a natural Vitamin B-complex, i.e., Panmol-B-complex - B1 (2.93 mg), B2 (3.98 mg), B3 (29.85 mg), B5 (10.95 mg), B6 (3.38 mg), B7 (0.108 mg), B9 (0.69 mg), B12 (8.85 µg) daily each morning for 6 weeks.The study finished after the second wash-out period for another 6 weeks.
  Interventions: Dietary Supplement: Synthetic Vitamin B-Complex

INTERVENTIONS:
Dietary Supplement: Natural Panmol-B-Complex — Natural Panmol-B-Complex: B1 (2.93 mg), B2 (3.98 mg), B3 (29.85 mg), B5 (10.95 mg), B6 (3.38 mg), B7 (0.108 mg), B9 (0.69 mg), B12 (8.85 µg) - Synthetic Vitamin B-Complex - B1 (2.93 mg), B2 (3.98 mg), B3 (29.85 mg), B5 (10.95 mg), B6 (3.38 mg), B7 (0.108 mg), B9 (0.69 mg), B12 (8.85 µg)
  Arms: Natural Panmol-B-Complex first, then synthetic Vitamin B-complex
Dietary Supplement: Synthetic Vitamin B-Complex — Synthetic Vitamin B-Complex: B1 (2.93 mg), B2 (3.98 mg), B3 (29.85 mg), B5 (10.95 mg), B6 (3.38 mg), B7 (0.108 mg), B9 (0.69 mg), B12 (8.85µg) - Natural Panmol-B-Complex: B1 (2.93 mg), B2 (3.98 mg), B3 (29.85 mg), B5 (10.95 mg), B6 (3.38 mg), B7 (0.108 mg), B9 (0.69 mg), B12 (8.85 µg)
  Arms: Synthetic Vitamin B-complex first, then Natural Panmol-B-Complex

SUMMARY:
In a cross-over study the investigators evaluate the effects of natural (Panmol-B-Complex) (Pan [Greek] = all; moles [Latin] = molecules/particles - brand name) versus synthetic vitamin B complexes to identify the bioavailability of distinct vitamins as well as long-term effects. The primary hypothesis for this study: "Natural Vitamin B-complexes are as effective as synthetic Vitamin B-complexes or better." For this reason 30 subjects (18 to 65y; BMI >19 to <29) were recruited for this study. The study population was divided into 2 groups of each 15 subjects in a cross-over trial. Vitamin supplementation consisted of Thiamine (2.93 mg), Riboflavin (3.98 mg), Niacin (29.85 mg), Pantothenic acid (10.95 mg), Pyridoxine (3.38 mg), Biotin (0.108 mg), Folic acid (0.69 mg) and Cobalamin (8.85 µg) per day in both groups. Blood samples are taken at baseline - 1.5h after vitamin supplementation - 4h - 7h - 6 weeks - wash out phase I (2 weeks); start cross-over: baseline - 1.5h after vitamin supplementation - 4h - 7h - 6 weeks - washout phase II (6 weeks). In case of main target criteria Thiamin, Riboflavin, Pyridoxine, Folic acid and Cobalamin were measured in serum as well as total peroxides (µmol/L), peroxidase-activity (U/L), total antioxidant status (mmol/L) and polyphenols (mmol/L).

DETAILED DESCRIPTION:
Design:

Monocentric double-blind experiment

Scientific background:

Vitamin B-complex is water-soluble and essential for humans. Vitamin B deficiency is associated with neurologic diseases, heart insufficiency, diminished hormone production and maldigestion. Due to the fact that literature search did not reveal distinct information about natural versus synthetic Vitamin B-complexes this study was initiated to investigate bioavailability and long-term effects of natural Vitamin B-complexes in comparison to synthetic Vitamin B-complexes.

Vitamin B complex was filled in hydroxypropylmethylcellulose capsules (size 0, ivory-coloured). Daily dose = 3 capsules in the morning with 250ml water.

Blinding/Randomization:

The person in charge for manufacturing and blinding arranged an identical packaging of both verum as well as synthetic Vitamin B-complex. Each package consists of 126 capsules per subject and period. Each product was tagged with the subject-number and period (period I and period II).

Study-subjects were blinded by the person in charge for randomization through a sealed envelope. The allocation was in the relation of 1:1 between group A (verum in period I and synthetic Vitamin B-complex in period II) and group B (synthetic Vitamin B-complex in period I and verum in period II). The ultimate subject list was forwarded to the person in charge for randomization after the run-in phase.

Method:

Blood sampling:

Blood (max. 20ml) was collected in a seated position from an antecubital vein.

Time schedule:

Run-in-phase: 3 weeks (no supplementation) Determination of inclusion criteria, nutrition advice, randomization.

Phase I: 6 weeks (supplementation) Group A - natural Vitamin B-complex supplementation every day Group B - synthetic Vitamin B-complex supplementation every day

Blood sampling:

First day:

Fasting value (basic) - Vitamin B-complex supplementation - After 1.5 hours After 4 hours After 7 hours

End of first supplementation:

After 6 weeks

Wash-out period: 2 weeks (without supplementation)

Phase II: 6 weeks (supplementation) Group A - synthetic Vitamin B-complex supplementation every day Group B - natural Vitamin B-complex supplementation every day

Blood sampling:

First day:

Fasting value (basic) - Vitamin B-complex supplementation - After 1.5 hours After 4 hours After 7 hours

End of second supplementation:

After 6 weeks

Wash-out period II: 6 weeks (without supplementation) Final exam - last blood sampling

Drop-out-criteria:

Drawback Compliance (<80% of Vitamin B-complexes) Supplementation of Vitamin B-complexes during run-in-phase or wash-out periods

Primary-target parameters:

Serum concentrations for vitamins B1, B2, B6, B9 and B12

Secondary-target biomarkers:

Serum concentrations for Total antioxidants, total peroxides, peroxidase-activity, polyphenols and homocysteine.

Biometry:

Comparison of interventions in a cross-over approach descriptive and exploratory.

Group comparison: Parametric and non-parametric cross-over comparison Gaussian distribution - (Kolmogorov-Smirnov-test with Lilliefors-significances, alpha =10%).

Effect size: Two-sided 95%-confidence intervals

Analysis:

Intent-to-treat-analysis Per-protocol-analysis Full analysis set

Vitamin B and Homocysteine analysis was done in a routine laboratory. Antioxidants (TAC), peroxidase-activity (EPA), peroxides (TOC) and polyphenols (PPm) were measured by the use of commercially available microtitre assays at a wavelength of 450 vs. 620 nm. In case of PPm a wavelength of 766nm was used.

Implausible values will be scored as missing values. Missing values are not substituted.

Presentation of results:

Minimum-Median-Quartiles-Maximum-Mean-Standard deviation. Box Plots, Bar graph, tables.

ELIGIBILITY:
Inclusion Criteria:

* Male and female
* 18-65 y
* Healthy

Exclusion Criteria:

* Cholesterol >240mg/dl
* Study inclusion in the past 2 months
* Pregnancy and lactation period
* Clinical diagnosis of chronic infections
* Ingestion of trace elements, vitamin- and fatty acid supplements in the past 3 months
* Clinical diagnosis of cardiovascular disease
* Clinical diagnosis of cancer
* Clinical diagnosis of psychotic diseases
* Insulin dependent diabetes
* Clinical diagnosis of autoimmune diseases
* Maldigestion/Malabsorption
* Veganes cuisine
* > 1 Beer/day

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-05-08 (Actual); Primary Completion 2017-10-03 (Actual); Study Completion 2017-11-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Wonisch Willibald, Graz, Styria, Austria

REFERENCES:
- [Result] Lindschinger M, Tatzber F, Schimetta W, Schmid I, Lindschinger B, Cvirn G, Stanger O, Lamont E, Wonisch W. A Randomized Pilot Trial to Evaluate the Bioavailability of Natural versus Synthetic Vitamin B Complexes in Healthy Humans and Their Effects on Homocysteine, Oxidative Stress, and Antioxidant Levels. Oxid Med Cell Longev. 2019 Dec 12;2019:6082613. doi: 10.1155/2019/6082613. eCollection 2019. PMID 31915511
- [Result] Lindschinger M, Tatzber F, Schimetta W, Schmid I, Lindschinger B, Cvirn G, Fuchs N, Markolin G, Lamont E, Wonisch W. [Bioavailability of natural versus synthetic B vitamins and their effects on metabolic processes]. MMW Fortschr Med. 2020 Mar;162(Suppl 4):17-27. doi: 10.1007/s15006-020-0230-4. Epub 2020 Mar 19. German. PMID 32189314

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 36 subjects were screened for eligibility at an Outpatient Clinic in Laßnitzhöhe, Styria, Austria
Pre-assignment Details: Of 36 enrolled participants, 30 met inclusion criteria and were randomized to treatment, i.e., to receive a natural (n=15) or synthetic vitamin B complex (n=15) after a 3 weeks run-in phase.
Groups:
- Natural Panmol-B-Complex First, Then Synthetic Vitamin B-complex: Participants first received Panmol-B-Complex: B1 (2.93 mg), B2 (3.98 mg), B3 (29.85 mg), B5 (10.95 mg), B6 (3.38 mg), B7 (0.108 mg), B9 (0.69 mg), B12 (8.85µg) each morning for 6 weeks. After a washout period of 2 weeks, they then received Synthetic Vitamin B-complex: B1 (2.93 mg), B2 (3.98 mg), B3 (29.85 mg), B5 (10.95 mg), B6 (3.38 mg), B7 (0.108 mg), B9 (0.69 mg), B12 (8.85 µg) each morning for 6 weeks.
- Synthetic Vitamin B-complex First, Then Natural Panmol-B-Complex: Participants first received Synthetic Vitamin B-Complex: B1 (2.93 mg), B2 (3.98 mg), B3 (29.85 mg), B5 (10.95 mg), B6 (3.38 mg), B7 (0.108 mg), B9 (0.69 mg), B12 (8.85 µg) each morning for 6 weeks. After a washout period of 2 weeks, they then received Natural Panmol-B-Complex: B1 (2.93 mg), B2 (3.98 mg), B3 (29.85 mg), B5 (10.95 mg), B6 (3.38 mg), B7 (0.108 mg), B9 (0.69 mg), B12 (8.85 µg) each morning for 6 weeks.
Period: First Intervention (6 Weeks)
Arm/Group | Natural Panmol-B-Complex First, Then Synthetic Vitamin B-complex | Synthetic Vitamin B-complex First, Then Natural Panmol-B-Complex
Started | 15 | 15
Completed | 14 | 15
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0
Period: Washout (2 Weeks)
Arm/Group | Natural Panmol-B-Complex First, Then Synthetic Vitamin B-complex | Synthetic Vitamin B-complex First, Then Natural Panmol-B-Complex
Started | 14 | 15
Completed | 14 | 15
Not Completed | 0 | 0
Period: Second Intervention (6 Weeks)
Arm/Group | Natural Panmol-B-Complex First, Then Synthetic Vitamin B-complex | Synthetic Vitamin B-complex First, Then Natural Panmol-B-Complex
Started | 14 | 15
Completed | 14 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Natural Panmol-B-Complex First, Then Synthetic Vitamin B-complex: Participants first received a natural vitamin B complex i.e. Panmol-B-Complex - B1 (2.93 mg), B2 (3.98 mg), B3 (29.85 mg), B5 (10.95 mg), B6 (3.38mg), B7 (0.108 mg), B9 (0.69 mg), B12 (8.85 µg) daily each morning for 6 weeks. After a wash-out period of 2 weeks, they then received a synthetic vitamin B-complex - B1 (2.93 mg), B2 (3.98 mg), B3 (29.85 mg), B5 (10.95 mg), B6 (3.38 mg), B7 (0.108 mg), B9 (0.69 mg), B12 (8.85 µg) daily each morning for 6 weeks. The study finished after the second wash-out period for another 6 weeks.
- Synthetic Vitamin B-complex First, Then Natural Panmol-B-Complex: Participants first received a synthetic vitamin B complex i.e. B1 (2.93 mg), B2 (3.98 mg), B3 (29.85 mg), B5 (10.95 mg), B6 (3.38 mg), B7 (0.108 mg), B9 (0.69 mg), B12 (8.85 µg) daily each morning for 6 weeks. After a wash-out period of 2 weeks, they then received a natural vitamin B-complex i.e. Panmol-B-Complex - B1 (2.93 mg), B2 (3.98 mg), B3 (29.85 mg), B5 (10.95 mg), B6 (3.38 mg), B7 (0.108 mg), B9 (0.69 mg), B12 (8.85 µg) daily each morning for 6 weeks. The study finished after the second wash-out period for another 6 weeks.
- Total: Total of all reporting groups
Arm/Group | Natural Panmol-B-Complex First, Then Synthetic Vitamin B-complex | Synthetic Vitamin B-complex First, Then Natural Panmol-B-Complex | Total
Number analyzed (Participants) | 14 | 15 | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 15 | 29
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 10 | 21
  Male | 3 | 5 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Ethnicity (NIH/OMB): Hispanic or Latino | 0 | 0 | 0
  Ethnicity (NIH/OMB): Not Hispanic or Latino | 14 | 15 | 29
  Ethnicity (NIH/OMB): Unknown or Not Reported | 0 | 0 | 0
  Race (NIH/OMB): Hispanic or Latino | 0 | 0 | 0
  Race (NIH/OMB): Not Hispanic or Latino | 14 | 15 | 29
  Race (NIH/OMB): Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Austria | 14 | 15 | 29

OUTCOME MEASURES:

1. Primary Outcome: Serum Thiamine
Description: Serum Thiamine in microgram per liter Minimum: 36 Maximum: 98
Time Frame: 20 weeks
Measure: Mean (Standard Deviation); unit: "µg/L"
Groups:
- Panmol-B-Complex: Participants first received a natural vitamin B complex i.e. Panmol-B-Complex - B1 (2.93 mg), B2 (3.98 mg), B3 (29.85 mg), B5 (10.95 mg), B6 (3.38 mg), B7 (0.108 mg), B9 (0.69 mg), B12 (8.85 µg) daily each morning for 6 weeks. After a wash-out period of 2 weeks, they then received a synthetic vitamin B-complex - B1 (2.93 mg), B2 (3.98 mg), B3 (29.85 mg), B5 (10.95 mg), B6 (3.38 mg), B7 (0.108 mg), B9 (0.69 mg), B12 (8.85 µg) daily each morning for 6 weeks. The study finished after the second wash-out period for another 6 weeks.
- Synthetic Vitamin B-complex: Participants first received a synthetic vitamin B complex i.e. B1 (2.93 mg), B2 (3.98 mg), B3 (29.85 mg), B5 (10.95 mg), B6 (3.38 mg), B7 (0.108 mg), B9 (0.69 mg), B12 (8.85 µg) daily each morning for 6 weeks. After a wash-out period of 2 weeks, they then received a natural vitamin B-complex i.e. Panmol-B-Complex - B1 (2.93 mg), B2 (3.98 mg), B3 (29.85 mg), B5 (10.95 mg), B6 (3.38 mg), B7 (0.108 mg), B9 (0.69 mg), B12 (8.85 µg) daily each morning for 6 weeks. The study finished after the second wash-out period for another 6 weeks.
Arm/Group | Panmol-B-Complex | Synthetic Vitamin B-complex
Number analyzed (Participants) | 14 | 15
"µg/L"
  Baseline | 50.21 (8.07) | 48.33 (6.51)
  1.5 hours | 51.21 (8.11) | 50.60 (8.72)
  4 hours | 53.57 (7.45) | 51.07 (7.20)
  7 hours | 52.00 (7.06) | 50.27 (8.74)
  6 weeks | 61.86 (9.81) | 61.33 (9.39)
  8 weeks | 70.14 (12.04) | 72.33 (10.75)
  8 weeks - 1.5 hours | 70.21 (8.94) | 69.13 (9.77)
  8 weeks - 4 hours | 64.71 (8.91) | 65.13 (10.95)
  8 weeks - 7 hours | 64.64 (8.14) | 64.20 (7.27)
  14 weeks | 58.86 (10.50) | 61.60 (9.91)
  20 weeks | 58.43 (10.52) | 59.20 (9.70)

2. Primary Outcome: Serum Riboflavin
Description: Serum Riboflavin in microgram per liter Minimum: 190 Maximum: 341
Time Frame: 20 weeks
Measure: Mean (Standard Deviation); unit: "µg/L"
Arm/Group | Panmol-B-Complex | Synthetic Vitamin B-complex
Number analyzed (Participants) | 14 | 15
"µg/L"
  Baseline | 231.93 (10.97) | 234.67 (21.87)
  1.5 hours | 233.86 (17.91) | 245.60 (21.88)
  4 hours | 240.36 (18.14) | 254.33 (27.63)
  7 hours | 247.21 (20.08) | 252.87 (27.03)
  6 weeks | 264.21 (17.62) | 265.00 (28.83)
  8 weeks | 232.29 (13.29) | 238.73 (14.18)
  8 weeks - 1.5 hours | 230.43 (9.72) | 233.27 (21.63)
  8 weeks - 4 hours | 237.36 (13.11) | 243.20 (15.42)
  8 weeks - 7 hours | 244.64 (8.11) | 250.13 (14.71)
  14 weeks | 258.14 (15.68) | 271.07 (20.66)
  20 weeks | 257.93 (12.75) | 274.67 (28.30)

3. Primary Outcome: Serum Pyridoxine
Description: Serum Pyridoxine in microgram per liter Minimum: 3.8 Maximum: 161.8
Time Frame: 20 weeks
Measure: Mean (Standard Deviation); unit: "µg/L"
Arm/Group | Panmol-B-Complex | Synthetic Vitamin B-complex
Number analyzed (Participants) | 14 | 15
"µg/L"
  Baseline | 23.11 (13.18) | 24.31 (25.80)
  1.5 hours | 35.45 (20.64) | 33.80 (29.23)
  4 hours | 32.96 (17.95) | 33.28 (28.81)
  7 hours | 36.66 (21.89) | 36.59 (25.83)
  6 weeks | 46.44 (20.10) | 48.94 (39.41)
  8 weeks | 29.23 (26.99) | 26.99 (33.38)
  8 weeks - 1.5 hours | 33.79 (20.71) | 36.93 (36.49)
  8 weeks - 4 hours | 39.14 (28.20) | 35.76 (32.58)
  8 weeks - 7 hours | 42.93 (27.35) | 40.41 (39.87)
  14 weeks | 42.24 (20.64) | 39.97 (26.30)
  20 weeks | 28.38 (26.26) | 21.39 (26.69)

4. Primary Outcome: Serum Folic Acid
Description: Serum Folic acid in nanogram per liter Minimum: 2.20 Maximum: 58.10
Time Frame: 20 weeks
Measure: Mean (Standard Deviation); unit: "ng/L"
Arm/Group | Panmol-B-Complex | Synthetic Vitamin B-complex
Number analyzed (Participants) | 14 | 15
"ng/L"
  Baseline | 7.45 (3.29) | 6.00 (2.79)
  1.5 hours | 25.21 (10.17) | 20.75 (8.32)
  4 hours | 12.87 (4.67) | 10.93 (2.96)
  7 hours | 10.38 (3.54) | 8.23 (2.62)
  6 weeks | 13.86 (2.77) | 15.18 (4.96)
  8 weeks | 11.04 (2.80) | 10.43 (3.04)
  8 weeks - 1.5 hours | 26.63 (10.52) | 31.87 (14.51)
  8 weeks - 4 hours | 16.39 (6.82) | 14.43 (2.29)
  8 weeks - 7 hours | 12.63 (2.48) | 12.19 (2.10)
  14 weeks | 18.59 (11.64) | 18.70 (14.42)
  20 weeks | 10.46 (2.33) | 9.93 (3.36)

5. Primary Outcome: Serum Cobalamin
Description: Serum Cobalamin in picogram per liter Minimum: 159 Maximum: 1230
Time Frame: 20 weeks
Measure: Mean (Standard Deviation); unit: "pg/L"
Arm/Group | Panmol-B-Complex | Synthetic Vitamin B-complex
Number analyzed (Participants) | 14 | 15
"pg/L"
  Baseline | 381.71 (112.73) | 440.47 (246.82)
  1.5 hours | 387.79 (122.48) | 453.67 (235.70)
  4 hours | 384.50 (105.92) | 447.00 (210.03)
  7 hours | 388.57 (116.72) | 442.27 (213.16)
  6 weeks | 442.36 (142.74) | 506.47 (166.44)
  8 weeks | 414.79 (125.67) | 450.33 (143.61)
  8 weeks - 1.5 hours | 414.57 (132.69) | 454.07 (141.05)
  8 weeks - 4 hours | 389.21 (115.06) | 432.07 (131.89)
  8 weeks - 7 hours | 404.93 (111.60) | 453.13 (129.37)
  14 weeks | 483.57 (139.02) | 564.27 (170.41)
  20 weeks | 421.07 (134.95) | 494.80 (176.79)

6. Secondary Outcome: Serum Total Peroxides
Description: Serum Total peroxides in micromol per liter Minimum: 23 Maximum: 443
Time Frame: 20 weeks
Measure: Mean (Standard Deviation); unit: "µM/L"
Arm/Group | Panmol-B-Complex | Synthetic Vitamin B-complex
Number analyzed (Participants) | 14 | 15
"µM/L"
  Baseline | 100.00 (46.17) | 111.17 (96.01)
  1.5 hours | 101.64 (38.65) | 112.67 (88.23)
  4 hours | 132.55 (43.72) | 137.08 (95.05)
  7 hours | 122.18 (46.42) | 132.75 (108.81)
  6 weeks | 97.36 (39.69) | 99.58 (31.84)
  8 weeks | 79.27 (25.86) | 71.25 (25.69)
  8 weeks - 1.5 hours | 97.27 (22.36) | 86.92 (25.04)
  8 weeks - 4 hours | 99.91 (23.28) | 92.50 (24.99)
  8 weeks - 7 hours | 89.18 (20.04) | 90.17 (27.33)
  14 weeks | 102.91 (23.78) | 115.83 (64.46)
  20 weeks | 104.91 (39.91) | 116.33 (105.86)

7. Secondary Outcome: Serum Total Antioxidant Capacity
Description: Serum total antioxidant capacity in millimole per liter Minimum: 0.31 Maximum: 2.45
Time Frame: 20 weeks
Measure: Mean (Standard Deviation); unit: "mM/L"
Arm/Group | Panmol-B-Complex | Synthetic Vitamin B-complex
Number analyzed (Participants) | 14 | 15
"mM/L"
  Baseline | 1.15 (0.43) | 1.45 (0.23)
  1.5 hours | 1.27 (0.31) | 1.24 (0.24)
  4 hours | 1.13 (0.33) | 1.23 (0.34)
  7 hours | 1.22 (0.44) | 1.39 (0.40)
  6 weeks | 1.45 (0.38) | 1.54 (0.22)
  8 weeks | 1.20 (0.22) | 1.31 (0.29)
  8 weeks - 1.5 hours | 1.68 (0.52) | 1.86 (0.30)
  8 weeks - 4 hours | 1.14 (0.38) | 1.30 (0.34)
  8 weeks - 7 hours | 1.38 (0.32) | 1.18 (0.57)
  14 weeks | 1.46 (0.32) | 1.48 (0.33)
  20 weeks | 1.34 (0.28) | 1.47 (0.38)

8. Secondary Outcome: Serum Endogenous Peroxidase-activity
Description: Serum endogenous peroxidase-activity in milliunits per milliliter Minimum: 0.79 Maximum: 9.87
Time Frame: 20 weeks
Measure: Mean (Standard Deviation); unit: "mU/mL"
Arm/Group | Panmol-B-Complex | Synthetic Vitamin B-complex
Number analyzed (Participants) | 14 | 15
"mU/mL"
  Baseline | 3.37 (1.74) | 3.07 (1.09)
  1.5 hours | 3.35 (1.49) | 3.90 (2.03)
  4 hours | 4.37 (1.26) | 4.22 (1.03)
  7 hours | 5.31 (1.13) | 4.84 (0.93)
  6 weeks | 4.36 (0.83) | 4.34 (0.55)
  8 weeks | 6.05 (1.82) | 5.15 (1.24)
  8 weeks - 1.5 hours | 3.97 (1.62) | 3.60 (1.03)
  8 weeks - 4 hours | 3.99 (1.12) | 3.93 (1.41)
  8 weeks - 7 hours | 4.35 (1.30) | 5.48 (1.74)
  14 weeks | 3.89 (1.53) | 4.95 (2.01)
  20 weeks | 3.04 (1.34) | 2.96 (1.14)

9. Secondary Outcome: Serum Polyphenols
Description: Serum Polyphenols in millimole per liter Minimum: 7.45 Maximum: 10.91
Time Frame: 20 weeks
Measure: Mean (Standard Deviation); unit: "mM/L"
Arm/Group | Panmol-B-Complex | Synthetic Vitamin B-complex
Number analyzed (Participants) | 14 | 15
"mM/L"
  Baseline | 9.88 (0.34) | 9.57 (0.34)
  1.5 hours | 9.73 (0.45) | 9.77 (0.67)
  4 hours | 9.97 (0.38) | 9.81 (0.45)
  7 hours | 9.72 (0.31) | 9.54 (0.43)
  6 weeks | 9.49 (0.35) | 9.46 (0.41)
  8 weeks | 9.73 (0.29) | 9.54 (0.53)
  8 weeks - 1.5 hours | 8.87 (0.66) | 8.71 (0.42)
  8 weeks - 4 hours | 8.25 (0.70) | 8.18 (0.70)
  8 weeks - 7 hours | 8.68 (0.35) | 8.57 (0.40)
  14 weeks | 8.72 (0.52) | 8.82 (0.44)
  20 weeks | 9.67 (0.34) | 9.46 (0.64)

10. Secondary Outcome: Total Homocysteine
Description: Total Homocysteine in Micromole Minimum: 4.00 Maximum: 40.40
Time Frame: 20 weeks
Measure: Mean (Standard Deviation); unit: "µM"
Arm/Group | Panmol-B-Complex | Synthetic Vitamin B-complex
Number analyzed (Participants) | 14 | 15
"µM"
  Baseline | 8.89 (1.99) | 11.49 (7.57)
  1.5 hours | 8.96 (2.32) | 11.89 (8.20)
  4 hours | 8.68 (1.98) | 11.38 (8.01)
  7 hours | 8.91 (2.03) | 11.31 (7.89)
  6 weeks | 7.76 (1.43) | 7.85 (1.89)
  8 weeks | 7.89 (1.58) | 8.16 (1.58)
  8 weeks - 1.5 hours | 7.91 (1.47) | 7.97 (1.45)
  8 weeks - 4 hours | 7.34 (1.45) | 7.39 (1.31)
  8 weeks - 7 hours | 8.00 (1.70) | 8.13 (1.69)
  14 weeks | 7.01 (1.59) | 7.44 (1.55)
  20 weeks | 7.62 (2.03) | 7.95 (1.88)

ADVERSE EVENTS:
Time Frame: 6 months
Groups:
- Natural Panmol-B-Complex: Participants received a Natural Panmol-B-Complex - B1 (2.93 mg), B2 (3.98 mg), B3 (29.85 mg), B5 (10.95 mg), B6 (3.38 mg), B7 (0.108 mg), B9 (0.69 mg), B12 (8.85 µg) daily each morning for 6 weeks.
- Synthetic Vitamin-B-Complex: Participants received a Synthetic Vitamin-B-Complex consisting of - B1 (2.93 mg), B2 (3.98 mg), B3 (29.85 mg), B5 (10.95 mg), B6 (3.38 mg), B7 (0.108 mg), B9 (0.69 mg), B12 (8.85 µg) daily each morning for 6 weeks (matching the Natural Panmol-B-Complex).
Arm/Group | Natural Panmol-B-Complex | Synthetic Vitamin-B-Complex
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 1/30 | 0/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Natural Panmol-B-Complex (N=30) | Synthetic Vitamin-B-Complex (N=30)
Flush (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-04-13): https://cdn.clinicaltrials.gov/large-docs/55/NCT03444155/Prot_SAP_000.pdf